CLINICAL TRIAL: NCT04967768
Title: The Influence and Effects of the COVID-19 Pandemic on Orthopaedic Resident Training: a Nationwide Cross-sectional Survey in Turkey
Brief Title: The Influence and Effects of the COVID-19 Pandemic on Orthopaedic Resident Training
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Huseyin Bilgehan Cevik, MD, Assoc. Prof., Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: 99/12
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Educational Problems; Covid19; Burnout, Student; Depression
MeSH Terms: conditions — COVID-19; Burnout, Psychological; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire about impact of the COVID-19 pandemic on orthopaedic resident training — Answers were collected for the effects of the COVID-19 pandemic on the real-life experiences of orthopaedic residents

SUMMARY:
Orthopedic residents, like all other healthcare professionals, face unique challenges during the coronavirus disease 2019 (COVID-19). The rapid spread of COVID-19 has forced healthcare systems around the world to adapt. As in many other specialties, it has led to many changes in the training of orthopedic residents including restructuring of surgical training, a reduction in elective surgery cases, and re-assignment of residents to COVID-19-related clinical duties. As a result, the standard training curriculum has been interrupted and the number of surgical cases has decreased, limiting the ability of the residents to meet the range and number of patient follow-up and treatment requirements set by the Turkish Orthopedics and Traumatology Education Council (TOTEK).

The already stressful work environment of orthopedic residents has become more stressful and anxious with the COVID-19 pandemic.

There are no well-designed survey studies that have shown the impact of the COVID-19 pandemic on orthopedic resident education and well-being from the resident's perspective. Therefore, the purpose of this nationwide survey study was to document and analyze the effects of the COVID-19 pandemic on the real-life experiences of orthopedic residents in Turkey.

ELIGIBILITY:
Inclusion Criteria:

Volunteering to answer survey questions

Exclusion Criteria:

Incomplete answers to survey questions or refusing to participate in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Orthopedic Residents in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The impact of the COVID-19 pandemic on orthopaedic resident training | 30.12.2020 - 15.01.2021
  Descriptive data on perceptions of current status of orthopaedic residency training during the pandemic and impact of the pandemic on orthopaedic residency training.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided